CLINICAL TRIAL: NCT05167760
Title: Efficacy of Topical Apraclonidine for the Treatment of Ocular Synkinesis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The project never opened.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Benjamin Greene, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008023
Record Dates: First submitted 2021-11-22; First posted 2021-12-22 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Synkinesis; Facial Nerve Palsy
MeSH Terms: conditions — Synkinesis; Bell Palsy | interventions — apraclonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Participants will receive the study drug, apraclonidine, per its FDA-approved package labelling
  Interventions: Drug: Apraclonidine

INTERVENTIONS:
Drug: Apraclonidine — 1-2 drops per eye every 8 hours for 2 weeks
  Other Names: Iopidine

SUMMARY:
The purpose of this study is to determine efficacy of apraclonidine for patients with ocular synkinesis, who are seen in the UAB Facial Nerve Clinic.

DETAILED DESCRIPTION:
UAB has a large Facial Nerve Clinic that treats patients with acquired facial nerve palsies and the associated difficulties of swallowing/speaking, and visual field defects from ptosis (a drooping or falling of the upper eyelid) and synkinesis (unwanted contractions of the muscles of the face during attempted movement.). Commonly, patients will experience involuntary eyelid contraction with oral movements like smiling. For eyelid synkinesis causing significant aesthetic or functional difficulty, surgery or botox is often the first line treatment. However, not all patients desire this, and some are poor surgical candidates due to other comorbidities. Botox has been shown to work well for these patients, but can be only partially effective. In addition, patients experience a wearing off period between treatments.

Several eye drops are available for the medical treatment of ptosis, including apraclonidine and 0.1% oxymetazoline. Both are alpha 2 adrenergic agonists, which stimulates Mullers muscle, causing muscle contraction and upper eyelid lifting. In addition, apraclonidine has been shown to be beneficial in patients with blepharospasm in a pilot study by Vijayakumar et. al.

We hypothesize that patients with synkinesis, similar to patients with ptosis and blepharospasm, could have symptomatic improvement with apraclonidine use.

Our study will initially be a pilot study, designed similarly to the Vijayakumar study. If this shows improvement for these patients, our hope is to pursue a randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability to speak and comprehend English
* Ability to consent for themselves
* Diagnosis of synkinesis affecting eye movement

Exclusion Criteria:

* Age less than 18 years
* Unable to speak and comprehend English
* Unable to consent for themselves
* Diagnosis of congenital ptosis, Horner syndrome, myasthenia travis, mechanical ptosis
* Visual field loss from causes unrelated to facial nerve injury
* Currently receiving monoamine oxidase inhibitors
* Known hypersensitivity to apraclonidine or other components of the drug under study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in synkinesis symptoms | Baseline - 20 minutes after study drug administration
  A 30 second video clip will be taken prior to administration of the study drug to record the unwanted movements of the facial muscles around the eyes. Approximately 20 minutes after study drug administration, a second 30-second video clip will be taken. Video clips from all of the participants will be pooled together at the end of the study and given to two independent raters. The raters will use the Sunnybrook Facial Grading System to assess each video and rate improvement of synkinesis after administration of the study drug. The Sunnybrook Facial Grading System rates resting symmetry (a scale of 0-2), symmetry of voluntary movement (a scale of 1-5), and synkinesis (a scale of 0-3), and computes a composite score. The higher the composite score, the better - full range of movement is scored as 100 percent.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greene, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No